CLINICAL TRIAL: NCT00791128
Title: A Phase II Single-Center, Prospective, Open Label Study of Safety and Efficacy, of the GI Sleeve for Pre-Surgical Weight Loss, in Type II Diabetes Patients (Cohort 06-6B Only)
Brief Title: Study for Pre-Surgical Weight Loss in Type II Diabetes Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-6
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EndoBarrier GI Liner (Experimental): 22 patients were implanted with the GI Liner for a 52-week duration. Assessments were performed during the 6 months post-explant period.
  Interventions: Device: GI Liner

INTERVENTIONS:
Device: GI Liner — Medical device placed endoscopically in the duodenum, nutritional counseling
  Other Names: GI Endobarrier Liner

SUMMARY:
The purpose of this study is to determine whether the GI Sleeve is safe and effective in treating Type II diabetes patients

DETAILED DESCRIPTION:
Patients with obesity are at significantly greater risk of developing complications such as pulmonary dysfunction, diabetes, hypertension, and other co-morbid risks. NIH panel recommendations state that even a 10% short-weight loss would greatly reduce these risks. GI Dynamics' GI Sleeve represents a viable alternative to other short-term pre-surgical weight loss methods. GI Sleeve is a device that can be implanted and removed through minimal invasive endoscopic techniques. This endoscopic procedure brings potential benefits to patients in that it is minimally invasive, efficacious, and allows patients to recover faster with less morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* BMI 40 to 60
* Type II Diabetes
* Candidates for bariatric surgery

Exclusion Criteria:

Patients with

* hepatitis B or C
* gastroesophageal reflux disease (GERD)
* HIV Positive diagnosis
* pancreatitis
* conditions of gastrointestinal tract, such as ulcers or Crohn's
* an infection or who are H. Pylori positive

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Guimaraes Hourneaux de Moura, MD, Principal Investigator — Hospital das Clinicas, Sao Paulo
Locations (1):
- Dr. Eduardo Guimaraes Hourneauz de Moura, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] de Moura EG, Martins BC, Lopes GS, Orso IR, de Oliveira SL, Galvao Neto MP, Santo MA, Sakai P, Ramos AC, Garrido Junior AB, Mancini MC, Halpern A, Cecconello I. Metabolic improvements in obese type 2 diabetes subjects implanted for 1 year with an endoscopically deployed duodenal-jejunal bypass liner. Diabetes Technol Ther. 2012 Feb;14(2):183-9. doi: 10.1089/dia.2011.0152. Epub 2011 Sep 20. PMID 21932999

RESULTS

PARTICIPANT FLOW:
Groups:
- EndoBarrier: Subjects implanted with the EndoBarrier for up to 12 months.
Period: Overall Study
Arm/Group | EndoBarrier
Started | 22
Completed | 13
Not Completed | 9
Not completed — Adverse Event | 4
Not completed — Device migration | 2
Not completed — non-compliance by subject | 2
Not completed — abdominal tumor, unrelated to device | 1

BASELINE CHARACTERISTICS:
Groups:
- EndoBarrier Liner Device: Subjects implanted with the EndoBarrier for up to 12 months.
Arm/Group | EndoBarrier Liner Device
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 22
Baseline Weight [Mean (Standard Deviation); unit: kg] | 119.2 (22.87)
Percent of glycosylated hemoglobin [Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin] | 8.9 (1.66)

OUTCOME MEASURES:

1. Primary Outcome: % of Excess Weight Loss (EWL)
Description: Percent excess weight loss (EWL) was calculated using Body Mass Index (BMI25) method: BMI25=ideal weight in kg/(height in meters)2 Ideal weight in kg = 25 x (Height in meters2) Baseline Excess weight = total weight - ideal weight
  % EWL = (baseline excess weight - weight loss) x 100
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: % excess weight loss
Arm/Group | EndoBarrier
Number analyzed (Participants) | 13
% excess weight loss | 37.7 (13.6)

2. Secondary Outcome: HbA1c Values at 12 Months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: HbA1c (%)
Arm/Group | EndoBarrier
Number analyzed (Participants) | 13
HbA1c (%) | 6.6 (1.1)

ADVERSE EVENTS:
Arm/Group | EndoBarrier
Serious Adverse Events (participants affected / at risk) | 2/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier (N=22)
Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal neoplasm (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Supra-ventricular tachycardia (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EndoBarrier (N=22)
Abdominal distention (Gastrointestinal disorders) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 20 (64)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 12 (23)
Vomiting (Gastrointestinal disorders) | 14 (30)
Asthenia (General disorders) | 11 (11)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Procedural nausea (Injury, poisoning and procedural complications) | 10 (13)
Procedural vomiting (Injury, poisoning and procedural complications) | 8 (8)
Blood cholesterol increased (Investigations) | 4 (4)
Blood iron decreased (Investigations) | 3 (3)
High density lipoprotein decreased (Investigations) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (21)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 4 (6)
Anxiety (Psychiatric disorders) | 2 (2)
Panic reaction (Psychiatric disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No